CLINICAL TRIAL: NCT06085599
Title: The Effect of Progressive Relaxation Exercises on Pain and Kinesiophobia After Liver Transplantation
Brief Title: The Effect of Exercises on Pain and Kinesiophobia in Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gurkan KAPIKIRAN (Other)
Responsible Party: Sponsor-Investigator, Gurkan KAPIKIRAN, Assistant Professor, Malatya Turgut Ozal University
Organization: Malatya Turgut Ozal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021-07/21-KAEK-109
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Liver Transplantation
Keywords: Liver Transplantation; Progressive Relaxation Exercises; Pain; Pain level; Kinesiophobia
MeSH Terms: conditions — Pain; Kinesiophobia

STUDY DESIGN:
Intervention Model Description: This study was conducted as a randomised controlled study with experimental and control groups.
Who Masked: Participant, Investigator
Masking Description: Participants did not know which group they were in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive relaxation exercise group (Experimental): Sociodemographic information form, numerical pain scale and kinesiophobia scale were applied to the patients in the experimental group after liver transplantation. They were shown 15 minutes progressive relaxation exercises prepared by Mark Connelly and Jennifer Bickel on Youtube, and then the numerical pain scale and kinesiophobia scale were applied again.
  Interventions: Behavioral: Progressive relaxation exercises
- Control group (No Intervention): No application other than clinical protocols was performed in the follow-up of the patient. In the control group, sociodemographic information form, kinesiophobia scale and numerical pain scale were applied after liver transplantation. No intervention was made. Then, the kinesiophobia scale and numerical pain scale were applied again.

INTERVENTIONS:
Behavioral: Progressive relaxation exercises — The progressive muscle relaxation technique involves suggestive stretching and relaxation in sixteen different muscle groups of the body. This technique is based on tensing each muscle group for approximately 10 seconds and then abruptly releasing this tension.
  Arms: Progressive relaxation exercise group

SUMMARY:
Liver transplantation is a treatment method used in acute and chronic liver failure. Progressive Relaxation Exercises, which are non-pharmacological methods aimed at minimizing complications and improving the quality of life after liver transplantation, have been reported to have many benefits such as reducing acute and chronic pain, reducing fatigue and reducing muscle tension. Therefore, in this study, the effects of progressive relaxation exercises on pain and kinesiophobia in liver transplant patients were examined.

DETAILED DESCRIPTION:
Liver transplantation is a common treatment for acute and chronic liver failure, liver malignancy and complicated cirrhosis. Although life expectancy increases after liver transplantation, some undesirable problems such as rejection, cardiovascular risk factors, hypertension, infection and malignancy occur. Preferring non-pharmacological methods to minimise complications and improve quality of life accelerates the return of the individual to normal life. Progressive Relaxation Exercises, one of these methods, can activate the parasympathetic nervous system, blood pressure, heart and respiratory rate can be kept within clinically normal limits due to vasodilatation in the blood vessels in the peripheral area and oxygen requirement is reduced. PGE has been reported to have many benefits such as reducing the effects of anxiety and stress, reducing acute and chronic pain, nausea and vomiting, facilitating sleep, reducing fatigue, reducing respiration, blood pressure, heart rate and muscle tension. Therefore, in this study, the effects of progressive relaxation exercises on pain and kinesiophobia in liver transplant patients were examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who agreed to participate in the study,
* Patients undergoing Liver Transplantation
* Patients without a disabling psychiatric disorder

Exclusion Criteria:

* Patients under the age of 18 who do not agree to participate in the study.
* Those who have a psychiatric diagnosis that prevents communication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Pain Level | up to 24 hours liver transplant (0-1 day
  The pain levels of the patients were measured by means of the visual pain scale.
  [Time Frame: up to 24 hours post-surgery (0-1 day)]
Tampa Kinesiophobia Scale (TKS) | up to 24 hours liver transplant (0-1 day
  The kinesiophobia levels of the patients were evaluated postoperatively and 24 hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- İnonu Üniversitesi Turgut Özal tıp Merkezi Karaciğer Nakil Enstitüsü, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No